CLINICAL TRIAL: NCT03241758
Title: Valuation Of Vascular Changes And Their Impact On Erectile Function By Penile Doppler Ultrasound And Analysis Of The Quality Of Life Of Patients Undergoing Laparoscopic Radical Prostatectomy
Brief Title: Vascular Changes Of Patients Undergoing Laparoscopic Radical Prostatectomy
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Jesus Muñoz-Rodriguez, Medical Doctor, Corporacion Parc Tauli
Other Study IDs: RadicalDoppler
Record Dates: First submitted 2017-08-03; First posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Prostatic Neoplasms; Erectile Dysfunction Following Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group #1: Patients with prostate cancer who will undergo radical prostatectomy
  Interventions: Diagnostic Test: Doppler ultrasound

INTERVENTIONS:
Diagnostic Test: Doppler ultrasound — Basal Doppler ultrasound and Doppler ultrasound one year after radical prostatectomy

SUMMARY:
A study designed to evaluate vascular changes after radical laparoscopic prostatectomy using Doppler ultrasound and the impact of such changes on erectile function and quality of life of patients. The baseline study will be compared with the study one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with prostate cancer who underwent laparoscopic radical prostatectomy

Exclusion Criteria:

* Patients who were not interested in their sexual function and refused to perform this study
* Patients who required adjuvant or salvage treatment for their prostate cancer (radiation therapy, chemotherapy or androgen deprivation therapy) during follow-up.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients with prostate cancer who underwent laparoscopic radical prostatectomy
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2011-11-29 (Actual); Primary Completion 2017-08-02 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
Left and right Cavernous artery diameter | 1 year
  mm
Left and right Systolic velocity cavernous artery | 1 year
  cm/s
Left and right Diastolyc velocity cavernous artery | 1 year
  cm/s

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Muñoz-Rodriguez, MD, Principal Investigator — Corporació Sanitaria Parc Tauli

IPD SHARING:
Plan to Share IPD: No